CLINICAL TRIAL: NCT01650584
Title: Evaluation of Ocular Comfort With ISTA Tears vs Systane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S00231
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISTA Tears (Experimental): Sterile ophthalmic solution
  Interventions: Drug: ISTA Tears
- Systane (Active Comparator): Sterile ophthalmic solution
  Interventions: Drug: Systane

INTERVENTIONS:
Drug: ISTA Tears — sterile ophthalmic solution
  Arms: ISTA Tears
Drug: Systane — Sterile ophthalmic solution
  Arms: Systane

SUMMARY:
To assess the comfort preference of ISTA Tears vs Systane in patients with dry eye disease (DED)

ELIGIBILITY:
Inclusion Criteria:

* OSDI >12

Exclusion Criteria:

* Presence of any active ocular disease other than dry eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 35 participants who applied ISTA Tears to the right eye and Systane to the left eye (70 eyes total).
Units Other Than Participants: eyes
Groups:
- All Participants: Each participant has 2 eyes. There were 35 participants who applied ISTA Tears to the right eye and Systane to the left eye (70 eyes total).
Period: Overall Study
Arm/Group | All Participants
Started | 35; 70 eyes (Each participant received one of 2 treatments in each eye.)
ISTA Tears | 35; 35 eyes
Systane | 35; 35 eyes
Completed | 35; 70 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: There were 35 participants who applied ISTA Tears to the right eye and Systane to the left eye (70 eyes total). The protocol required that participants be least 18 years of age, male or female. Participant demographic information was not collected.
Units Other Than Participants: Eyes
Groups:
- All Participants Received Both ISTA Tears and Systane: ISTA Tears: sterile ophthalmic solution used in the right eye.
  Systane: Sterile ophthalmic solution used in the left eye.
Arm/Group | All Participants Received Both ISTA Tears and Systane
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 70
Age, Customized [Count of Participants; unit: Participants]
  At least 18 years of age | 35
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Both male or female | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Preference for One of the Treatments
Description: There were 35 participants who applied ISTA Tears to the right eye and Systane to the left eye (70 eyes total). Participants were asked to indicate which treatment they preferred, or if they preferred neither.
Time Frame: 30 days
Population: There were 35 participants who applied ISTA Tears to the right eye and Systane to the left eye (70 eyes total).
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 35
Participants
  ISTA Tears preferred | 23
  Neither preferred | 1
  Systane preferred | 11

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Participants Received Both ISTA Tears and Systane: ISTA Tears: sterile ophthalmic solution used in the right eye.
  Systane: Sterile ophthalmic solution used in the left eye.
Arm/Group | Participants Received Both ISTA Tears and Systane
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for detail.